CLINICAL TRIAL: NCT05691777
Title: Counirs: Study of Cortical Activation During Hand and Shoulder Movements - Contribution of fNIRS in Healthy Subjects
Brief Title: Study of Cortical Activation During Hand and Shoulder Movements in Healthy Subjects
Acronym: CouNirs
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Other Study IDs: CHRO-2020-04
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Healthy
Keywords: cortical activation; functional near-infrared spectroscopy; upper limb; motricity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy participants: right handed healthy participants aged between 18 and 40.
  Interventions: Device: Hand and shoulder task

INTERVENTIONS:
Device: Hand and shoulder task — Hand task: the participant is seated on a chair facing a table, both hands resting on the table. The participant is asked, for each block of 10 seconds, to perform flexion / extension movements of the fingers of the right hand at 0.5 Hz.
  Shoulder task: the participant is seated on a chair facing a table, both hands resting on the table. The participant is asked, for each block of 10 seconds, to perform alternating movement of abduction and adduction of the right shoulder at 0.5 Hz with the elbow flexed.

SUMMARY:
Characterization of cortical activation patterns during movements in healthy adults may help our understanding of how the injured brain works. Upper limb motor tasks are commonly used to assess impaired motor function and to predict recovery in individuals with neurological disorders such as stroke. This study aimed to explore cortical activation patterns associated with movements of the hand and shoulder using functional near-infrared spectroscopy (fNIRS). The investigators hypothesized that the activation pattern observed with fNIRS would differ for shoulder and hand movements. More specifically, the investigators hypothesized that the cerebral activation during hand movements would mainly involve the contralateral hemisphere, particularly the lateral part of primary motor cortex; whereas activation during shoulder movements would be more medial and more extensive than that of the hand.

DETAILED DESCRIPTION:
Stroke is a leading cause of chronic disability worldwide in adults. Upper extremity (hand and arm) impairments are especially prevalent after stroke and cause lasting disabilities. Functional reorganization of the motor cortex may occur in both the ipsilesional and contralesional hemispheres. Thus, knowledge of brain activation patterns during execution of a movement is important both for neuroscience and neurorehabilitation.

The use of brain imaging techniques for post-stroke follow-up is valuable for understanding the mechanisms of cerebral recovery. Functional Near-Infrared Spectroscopy (fNIRS) is a non-invasive technique that assesses neural activation through the measurement of cortical oxygenated and deoxygenated hemoglobin concentrations during motor tasks in a natural.

As remapping of the sensorimotor cortex after stroke with hand impairment can involve the territory of the elbow or shoulder, the investigators aimed to determine if the cortical activation of these regions (hand and shoulder) could be distinguished by fNIRS recordings in healthy subjects. The investigators hypothesized that the activation pattern observed with fNIRS would differ for shoulder and hand movements. More specifically, the investigators hypothesized that the cerebral activation during hand movements would mainly involve the contralateral hemisphere, particularly the lateral part of primary motor cortex; whereas activation during shoulder movements would be more medial and more extensive than that of the hand, involving the contralateral premotor region and supplementary motor cortex. If these three cortical regions could be distinguished by fNIRS, this technique could be used to measure spontaneous motor recovery and rehabilitation-induced recovery after stroke.

The investigations will be carried out by the principal investigator or by specialized technicians from the neurology functional exploration department.

Each acquisition has a duration of 920 seconds, it begins with a rest period of 120 seconds, which corresponds to the baseline.

For each condition the movements are performed at a frequency of 0.5 Hz which seems to be the optimal frequency for observing cortical activation using a metronome. Each movement is therefore performed 10 times per block.

The order of placing the various conditions will be balanced. Between periods of movement, the subject is in a resting position for 30 seconds.

The "movement" and "rest" instructions are given at the start of each phase.

The protocol has 2 conditions:

* Shoulder task
* Hand task

After recruiting the participants, the study investigator will check the inclusion and non-inclusion criteria.

On the day of the first acquisition, the subject will present to the neurology department at the time of his appointment.

Then the fNIRS acquisition headset (Brite 24) will be installed by a specialized technician and the procurement instructions will be given.

The acquisition is then carried out. The helmet is only removed at the end of the acquisition

ELIGIBILITY:
Inclusion Criteria:

* Age:18 to 40
* Right handed
* No neurological, rhumatological or cardiac disease
* Having social security coverage
* Having expressed his non-objection

Exclusion Criteria:

* Person under tutorship or curatorship
* Known allergy to components of the fNIRS device: neoprene
* Person with known vascular problems

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: right handed healthy subjects aged between 18 and 40
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2020-07-16 (Actual); Study Completion 2020-07-16 (Actual)

PRIMARY OUTCOMES:
Mean change in the concentration of oxyhemoglobin and deoxyhemoglobin during the task | Day 0
  Changes in the concentration of oxyhemoglobin and deoxyhemoglobin during the task measured with fNIRS device

CONTACTS AND LOCATIONS:
Overall Officials: Julien BONNAL, Principal Investigator — CHR d'Orléans
Locations (1):
- CHR Orléans, Orléans, France

REFERENCES:
- [Background] Nudo RJ, Milliken GW. Reorganization of movement representations in primary motor cortex following focal ischemic infarcts in adult squirrel monkeys. J Neurophysiol. 1996 May;75(5):2144-9. doi: 10.1152/jn.1996.75.5.2144. PMID 8734610
- [Background] Carrera E, Jones PS, Morris RS, Alawneh J, Hong YT, Aigbirhio FI, Fryer TD, Carpenter TA, Warburton EA, Baron JC. Is neural activation within the rescued penumbra impeded by selective neuronal loss? Brain. 2013 Jun;136(Pt 6):1816-29. doi: 10.1093/brain/awt112. Epub 2013 May 16. PMID 23682070
- [Background] Csipo T, Mukli P, Lipecz A, Tarantini S, Bahadli D, Abdulhussein O, Owens C, Kiss T, Balasubramanian P, Nyul-Toth A, Hand RA, Yabluchanska V, Sorond FA, Csiszar A, Ungvari Z, Yabluchanskiy A. Assessment of age-related decline of neurovascular coupling responses by functional near-infrared spectroscopy (fNIRS) in humans. Geroscience. 2019 Oct;41(5):495-509. doi: 10.1007/s11357-019-00122-x. Epub 2019 Nov 2. PMID 31676966
- [Background] Delorme M, Vergotte G, Perrey S, Froger J, Laffont I. Time course of sensorimotor cortex reorganization during upper extremity task accompanying motor recovery early after stroke: An fNIRS study. Restor Neurol Neurosci. 2019;37(3):207-218. doi: 10.3233/RNN-180877. PMID 31227675
- [Background] Kato J, Yamada T, Kawaguchi H, Matsuda K, Higo N. Functional near-infrared-spectroscopy-based measurement of changes in cortical activity in macaques during post-infarct recovery of manual dexterity. Sci Rep. 2020 Apr 15;10(1):6458. doi: 10.1038/s41598-020-63617-0. PMID 32296087
- [Background] Lee SH, Jin SH, An J. The difference in cortical activation pattern for complex motor skills: A functional near- infrared spectroscopy study. Sci Rep. 2019 Oct 1;9(1):14066. doi: 10.1038/s41598-019-50644-9. PMID 31575954
- [Background] Yang CL, Lim SB, Peters S, Eng JJ. Cortical Activation During Shoulder and Finger Movements in Healthy Adults: A Functional Near-Infrared Spectroscopy (fNIRS) Study. Front Hum Neurosci. 2020 Jul 8;14:260. doi: 10.3389/fnhum.2020.00260. eCollection 2020. PMID 32733221
- [Background] Yeo SS, Chang PH, Jang SH. The cortical activation differences between proximal and distal joint movements of the upper extremities: a functional NIRS study. NeuroRehabilitation. 2013;32(4):861-6. doi: 10.3233/NRE-130910. PMID 23867412
- [Background] Pinti P, Tachtsidis I, Hamilton A, Hirsch J, Aichelburg C, Gilbert S, Burgess PW. The present and future use of functional near-infrared spectroscopy (fNIRS) for cognitive neuroscience. Ann N Y Acad Sci. 2020 Mar;1464(1):5-29. doi: 10.1111/nyas.13948. Epub 2018 Aug 7. PMID 30085354
- [Derived] Bonnal J, Ozsancak C, Monnet F, Valery A, Prieur F, Auzou P. Neural Substrates for Hand and Shoulder Movement in Healthy Adults: A Functional near Infrared Spectroscopy Study. Brain Topogr. 2023 Jul;36(4):447-458. doi: 10.1007/s10548-023-00972-x. Epub 2023 May 18. PMID 37202647